CLINICAL TRIAL: NCT00250120
Title: Pharmacology Study of Aerosolized Liposomal 9-Nitro-20 (S) - Camptothecin (L9NC)
Brief Title: Pharmacology Study of Aerosolized Liposomal
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Claire Verschraegen, MD; Principal Investigator, Universtiy of New Mexico - CRTC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1402C-T
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Lung Diseases; Cancer
Keywords: NSCLC; L9NC; Aerosolized Liposomal 9-Nitro-20 (S)-Camptothecin
MeSH Terms: conditions — Lung Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: L9NC: Liposomal 9-Nitro-20 (S)-Camptothecin — delivery mode: inhalation

SUMMARY:
To determine the overall response rate to liposomal 9-Nitro-20 (S)-Camptothecin (L9NC) administered by aerosolization in patients with non-small-cell lung cancer (any stage).

To determine toxicity profile of L9NC administered by aerosolization for 5 consecutive days per week X 8 weeks, every 10 weeks.

To perform a pharmacology study of L9NC in the plasma, and the lungs after aerosolization. A specific protocol will be written for this part.

DETAILED DESCRIPTION:
This is a single-arm, non-randomized Phase II trial of DLPC-9NC administered by aerosol 5 consecutive days per week for 8 weeks every 10 weeks.

Dose: 0.4 mg/ml of 9-NC in aerosol reservoir for 60 minutes (= daily dose of 0.52 mg/m2/day) per day X5 every week, X8 weeks, then observe for 2 weeks. One course = 10 weeks.

Patients that have a resectable lung cancer will only receive one course of treatment and will be operated on about two weeks after completing the 8-week course.

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in INST 1402C protocol
* Phase II Study of Aerosolized Liposomal-Nitro-20 (S)-Camptothecin (L9NC) in Patients with Advanced (NSCLC) Lung Cancer are eligible if their tumor is resectable with curative intent as determined by Dr. Reza Mehran.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-04; Primary Completion 2007-03 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Pathological examination of lung tissure | at surgery

CONTACTS AND LOCATIONS:
Overall Officials: Claire F Verschraegen, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States